CLINICAL TRIAL: NCT01157689
Title: The Routine Use of Coartem for Treatment of Symptomatic Children With Plasmodium Falciparum at the Bandim Health Centre
Brief Title: Artemether-Lumefantrine Effectiveness in Guinea-Bissau
Status: Completed | Type: Observational
Sponsor: Bandim Health Project (Other)
Responsible Party: Sponsor
Other Study IDs: AL-eff 2010
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Malaria
Keywords: malaria; children; Guinea-Bissau; artemether; lumefantrine; effectiveness
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Capillary blood samples for drug concentration analysis and for PCR for identifying the malaria parasites
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Coartem, chloroquine, quinine: All children with a positive malaria test will included. Results will be subanalysed acording to treatment given by routine health staff.

SUMMARY:
The routine treatment of children with antimalarials will be monitored. Children with a positive malaria film and/or a positive rapid diagnostic test (RDT) will be included in a follow-up study. The genetic basis of the parasites for developing resistance will be examined. In case of reappearance of parasites the child will be re-treated following the guidelines of the national malaria programme.

DETAILED DESCRIPTION:
Children from the Bandim area in Bissau who are seeking medical advice and who are recommended treatment for malaria in accordance with the current routines will be included as follows:

All children getting the clinical diagnosis of malaria will be registered and basic information collected. Of theses, children fulfilling the inclusion criteria will be included in a follow-up study.

The children included in the follow-up part of the study will be visited on day 7, day 14, day 21, day 28, day 35 and day 42. At each visit the condition of the child will be evaluated, a questionnaire will be filled in and a malaria film and approximately 100 µl blood on filter-paper (for PCR analysis in case of re-parasitaemia) will be taken. Furthermore, on day seven 100 μl blood on filter-paper will be taken for drug-analysis.

Children with parasitaemia detected by only one of the following methods will be excluded from the final analyses of the effectiveness: 1) malaria film, 2) RDT, and 3) PCR.

If the parents do not ensure that the children get the correct medication resulting in a high rate of recrudescence and/or a low drug-concentration on day seven the policy of the National Malaria Programme should be re-evaluated. If the health staff do not follow the guidelines of the National Malaria Programme the reasons why should be elucidated in order to ensure a better adherence.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed an anti-malarial at the Bandim Health Centre
* Having P. falciparum parasites in a thick film and/or a positive RDT
* The Bandim address is known (to enable follow up).

Exclusion Criteria:

* Children where the parents do not accept to participate in the study.
* Signs of severe malaria such as convulsion or severe anemia

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children diagnosed as having malaria at Bandim Health Center in Bissau. Of these all children with a positive malaria film and/or a positive rapid diagnostic test will be included in an observational follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-03 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
ACPR day 42 | day 42
  Malaria slides will be examined weekly during follow-up until day 42. The adequate clinical and parasitological cure rate will to calculated for day 42.

SECONDARY OUTCOMES:
ACPR day 28 | 28 days

OTHER OUTCOMES:
Side effects | During follow-up for 42 days
  All possible side effects will be recorded during the 42 day long follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandim Health Project, Bissau, Bissau Codex, Guinea-Bissau

REFERENCES:
- [Derived] Jovel IT, Kofoed PE, Rombo L, Rodrigues A, Ursing J. Temporal and seasonal changes of genetic polymorphisms associated with altered drug susceptibility to chloroquine, lumefantrine, and quinine in Guinea-Bissau between 2003 and 2012. Antimicrob Agents Chemother. 2015 Feb;59(2):872-9. doi: 10.1128/AAC.03554-14. Epub 2014 Nov 24. PMID 25421474